CLINICAL TRIAL: NCT03684759
Title: Pilot Feasibility Study for Cystic Fibrosis Sputum Validation for the Molecular Diagnosis of Respiratory Viral Infections
Brief Title: Sputum Validation for the Molecular Diagnosis of Respiratory Viral Infections in Cystic Fibrosis
Acronym: EXPIRE
Status: Completed | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: EXPIRE
Record Dates: First submitted 2018-09-21; First posted 2018-09-26 (Actual); Last update posted 2018-09-26 (Actual); Status verified 2018-09

CONDITIONS: Cystic Fibrosis; Respiratory Infection
Keywords: Expectoration; Cystic Fibrosis; Nasopharyngeal; Viral molecular diagnosis
MeSH Terms: conditions — Cystic Fibrosis; Respiratory Tract Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — respiratory samples were retained at -80°C
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this pilot study is to demonstrate the feasibility of viral biomolecular diagnosis in sputum compared to nasopharyngeal swab in cystic fibrosis acute respiratory infection.

DETAILED DESCRIPTION:
In cystic fibrosis (CF), patients face polymicrobial airway infections. Besides bacteria, viruses are now also considered as important agents in lung function deterioration. No strategy has been established on the optimal sampling for respiratory viral molecular diagnostic in CF. Nasopharyngeal swabs (NP) are recommended for respiratory viral screening in non-CF patients but are invasive and sometimes painful for patients. As sputa are non invasive and collected for bacterial monitoring in CF patients they could represent a convenient alternative to NP swabs.

This study's aim is to define whether viral screening give concordant results between sputa and NP swabs.

ELIGIBILITY:
Inclusion Criteria:

* Participant with Cystic Fibrosis
* Participant able to expectorate
* Participant with sign of acute respiratory infection

Exclusion Criteria:

* participant not able to expectorate
* patient refusing to participate

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: participant living with cystic fibrosis disease cared in french pediatric or adult CRCM
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2016-02-24 (Actual); Primary Completion 2017-02-06 (Actual); Study Completion 2017-02-06 (Actual)

PRIMARY OUTCOMES:
Concordance of viral type detected in both samples for each participant: sputum and nasopharyngeal swab | Day 1
  Comparison of per participant results of viral molecular detection in sputum and nasopharyngeal swab.
  Concordance=same virus(es) or no virus detected in both sample. no concordance=different viruses detected in each sample or virus(es) detected in only one sample and not in the other

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - CHU d'Angers, Angers
  - Centre de Perharidy, Roscoff
  - Hôpital Foch, Suresnes